CLINICAL TRIAL: NCT06084273
Title: Effectıveness Of Relaxation And Respiratory Exercise On Sleep Quality, Depressıon And Spasticity In Hemiplegic Stroke Patients: Prelimınary Findings
Brief Title: Investigation Of Two Different İnterventions İn Hemiplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derya Azim (Other)
Responsible Party: Sponsor-Investigator, Derya Azim, Assistant Professor, Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06.04/58
Record Dates: First submitted 2023-10-02; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Physiotherapy and Rehabilitation
Keywords: Depression; Exercise; Relaxation; Pain
MeSH Terms: conditions — Stroke; Depression; Motor Activity; Pain | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bobath Exercises (Experimental): Bobath Exercises
  Interventions: Other: Bobath Exercises
- Breathing Exercises,Breathing Exercises, Bobath Exercises (Experimental): Breathing Exercises,Breathing Exercises, Bobath Exercises
  Interventions: Other: Bobath Exercises; Other: Breathing Exercises,Breathing Exercises, Bobath Exercises

INTERVENTIONS:
Other: Bobath Exercises — The Bobath approach aims to enhance postural and neuromotor control goal-directedly, leading to functional improvement. Our study selected the Bobath 30 exercises from the fundamental exercises to create a program specific to the goal and targeting functionality.
  The ten Bobath exercises performed by all participants in the study are as follows: Bridging Exercise, Latissimus Stretch Exercise, Autoinhibition Exercise, Dorsiflexion Training, Sitting Balance Training, Upper Extremity Weight Shifting Exercise, Lower Extremity Weight Shifting Exercise, Oblique Abdominal Strengthening Exercise, Knee Control Training, and Walking Training.
Other: Breathing Exercises,Breathing Exercises, Bobath Exercises — The puckered lip breathing exercise aims to prevent the closure of the small airways by creating pressure during expiration. During the exercise, the individual is asked to follow these steps:
  1. Breathe calmly and slowly through the nose.
  2. Pucker the lips as if whistling or inflating a balloon.
  3. Exhale the breath with puckered lips. Relaxation exercises Progressive Muscle Relaxation Technique: Progressive muscle relaxation is one of the easiest methods to learn and apply, developed by Jacobson. It involves voluntarily tensing and relaxing large muscle groups regularly and sequentially. The participant was encouraged to wear comfortable clothing, breathe deeply, and exhale. The technique can be performed in a sitting or lying position. Music can be played to contribute to the participant's relaxation.
  Arms: Breathing Exercises,Breathing Exercises, Bobath Exercises

SUMMARY:
Background: Our study aims to determine the effect of relaxation and breathing exercises in addition to the treatment procedure on depression level, sleep quality, and spasticity in hemiplegic patients.

Methods: Thirty patients aged 40-70 years diagnosed with hemiplegia were included in the study. All patients received the same Bobath exercise three days a week for six weeks. Patients in Group 2 additionally received breathing and relaxation exercises. Sleep quality assessment by Pittsburgh Sleep Quality Index (PUKI), depression by Hospital Anxiety and Depression Scale (HADS), and spasticity by Modified Ashworth scale (MAS) were used. All assessments were made at baseline and six weeks after exercise treatments.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients who met the following inclusion criteria:
* having had a stroke at least six months ago,
* possessing adequate cognitive functions,
* having no pre-existing sleep problems before the disease,
* absence of emotional disturbance prior to the disease,
* voluntary participation in the study,
* no cardiovascular problems,
* having a score of 1, 1+, or two according to the modified Ashworth Scale

Exclusion Criteria:

* having a traumatic stroke caused by malignancy or other organic factors, alcohol or drug addiction,
* having a score of 3 or 4 according to the modified Ashworth Scale

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Sleep quality assessment | 30 min
  The subjective sleep questionnaire, the PUKI, is used to assess individuals' sleep quality, sleep duration, presence of sleep problems, and the severity of sleep problems over the past month.
Depression assessment | 30 min
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale developed to determine the risk, level, and severity of anxiety and depression in individuals
Spasticity assessment | 15 min
  Spasticity is a method used to determine the severity of spasticity. The assessment is based on the subjective rating of the resistance felt by the evaluator during the evaluation. It is divided into six degrees: 0 = Normal muscle tone, 1 = Slight increase in muscle tone with minimal resistance felt at the end of the range of motion, 1+ = Minimal resistance felt in less than half of the range of motion, 2 = more pronounced increase in muscle tone but affected parts can be moved without difficulty, 3 = Passive movement is complex and requires significant effort, with a noticeable increase in muscle tone, 4 = Affected parts are rigid in flexion and extension, with severe increase in tone.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No